CLINICAL TRIAL: NCT06049836
Title: Holographic Augmented Reality Versus Screen Visualisation of 3D Rendering Models for the Pre-operative Evaluation and Planning of Liver Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Collaborators: ICAR (Istituto di Calcolo e Reti ad Alte Prestazioni) - CNR (Consiglio Nazionale delle Ricerche) (Unknown)
Responsible Party: Principal Investigator, Gianluca Rompianesi, Assistant Professor of Surgery - MD, PhD, FEBS (HPB, Transplantation), Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FIICNRHoloLiver
Record Dates: First submitted 2023-09-08; First posted 2023-09-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hepatobiliary Neoplasm
Keywords: Liver surgery; Preoperative planning; 3D rendering; Augmented reality; Holograms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A analyses 15 patient cases 3D Hologram models (first stage) and after the washout period the same 15 patients cases (anonymised, renamed and shuffled) in liver 3D models on computer monitor visualisation (PDF) (second stage)
  Interventions: Other: Holograms; Other: PDF
- Group B (Experimental): Group B analyses 15 patient cases liver 3D models on computer monitor visualisation (PDF) (first stage) and after the washout period the same 15 patients cases (anonymised, renamed and shuffled) on 3D Hologram models (second stage)
  Interventions: Other: Holograms; Other: PDF

INTERVENTIONS:
Other: Holograms — Clinical decision making based on visualising liver 3D holographic augmented reality liver models
Other: PDF — Clinical decision making based on visualisation of 3D liver rendering on computer monitors on a PDF file

SUMMARY:
The goal of this trial is to compare the evaluation of 3D liver models visualised as holograms with HoloLens 2 and on digital PDF files in HPB surgical trainees.

The main questions it aims to answer are:

* Do the holographic models allow a superior accuracy in terms of anatomical evaluation and surgical planning?
* Is there any difference in terms of time consumed and Task Load Index? Participants will analyse cases through both modalities and answer a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* General Surgery Trainees with at least 6 months experience in HPB surgery

Exclusion Criteria:

* No informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic and planning accuracy | Immediately after completing the evaluation
  Correctly identify anatomy and appropriate surgical planning Residents' decision-making accuracy when reviewing patient data and 3D liver models using Holograms or on PDF, measured by comparing their performance.
  The measurement tool will be a questionnaire consisting of 11 questions, rate of correct answers will be recorded (e.g. 8/10 correct answers) and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Time consumed | Immediately after completing the evaluation
  Analyse the time spent for the evaluation of the cases and complete the questionnaire Assessed by total time needed to make decision for 15 patient cases in minutes
NASA Task Load Index | Immediately after completing the evaluation
  Analyse the NASA TLI score for each participant to evaluate the cases by conducting a subjective mental workload assessment rating performance across six dimensions to determine an overall workload rating:
  1. Mental demand - how much thinking, deciding, or calculating was required to perform the task.
  2. Physical demand - the amount and intensity of physical activity required to complete the task.
  3. Temporal demand - the amount of time pressure involved in completing the task.
  4. Effort - how hard does the participant have to work to maintain their level of performance?
  5. Performance - the level of success in completing the task.
  6. Frustration level - how insecure, discouraged, or secure or content the participant felt during the task.
  Each participant gives a rating for each subscale from 1 (low) to 20 (high) and the TLX will calculate the overall worklaod score between 0 and 100

CONTACTS AND LOCATIONS:
Overall Officials: Roberto I Troisi, MD PhD FEBS, Principal Investigator — Federico II University
Locations (1):
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD are to be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication